CLINICAL TRIAL: NCT01042470
Title: Pelvic Floor Study: Biomechanical Properties of the Female Pelvic Floor - Evaluation of Clinical, Mechanical, Sonographic and Histological Parameters
Brief Title: Pelvic Floor Study: Biomechanical Properties of the Female Pelvic Floor
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: David Scheiner (Other)
Collaborators: ETH Zurich (Switzerland) (Other); University of Zurich (Other)
Responsible Party: Sponsor-Investigator, David Scheiner, Oberarzt, University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: FHKUSZ11-2009
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolapse; pelvic floor dysfunction; biomechanics; aspiration device; connective tissue
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue (vaginal wall, urogenital diaphragm), whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- control group: female patients without pelvic organ prolapse, stage 0 or I (POP-Q)
- pelvic organ prolapse: female patients with pelvic organ prolapse stage II or higher (POP-Q)

SUMMARY:
Pelvic floor dysfunction in the form of pelvic organ prolapse or urinary and fecal incontinence is a sequela for some women who experience injuries during birth. It affects adult women of all ages. The life time risk for women by age of 80 years for undergoing surgical correction is shown to be 11.1 % , and 29 % of them will undergo re-operation for recurrences later on. Still, even today the biomechanics of the pelvic floor is not understood enough. The aim of our study is to investigate the biomechanical properties of the female pelvic floor, i.e. the vaginal wall, by means of clinical, sonomorphometric (ultrasound), histological and elastomechanical examinations. In principle, the elasto-mechanical properties of the vaginal wall will be examined by the new and innovative so called aspiration device, developed at the Eidgenoessische Technische Hochschule (ETH) Zurich, Switzerland. This tool generates a low-pressure of -25 mbar at the vaginal wall, aspirating it under visual control by aid of an integrated video camera and therefore allowing to measure the difference of its convexity under aspiration and at rest. In case of prolapse surgery, this allows us to take a biopsy of the measured vaginal wall and analyze it at the Institute of Anatomy at the University of Zurich-Irchel by means of histological (e.g. connective tissue, extracellular matrix) and molecular biological examination. With an increasing elderly population, more and more women will need surgery for pelvic organ prolapse. While effective in restoring anatomy, sometimes by aid of meshes made out of polypropylene, the functional outcomes and quality of life are not always restored satisfactorily. This interdisciplinary project intends to add a contribution to this for our patient still bothersome situation and to help to detect risk factors for developing pelvic floor dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* pre- and postmenopausal women
* with pelvic organ prolapse, i.e. cysto- or rectocele, uterine descensus
* postmenopausal women

Exclusion Criteria:

* age under 18 years
* pregnancy / lactation
* current gynaecologic malignancies
* current malignancies of the pelvic floor
* infections such as HPV
* treatment with steroids or methotrexate
* no informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: female patients who are referred to our university hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-01; Primary Completion 2015-06 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
normative values for the aspiration technique | one year
correlation of elasticity parameters with histology | one year

CONTACTS AND LOCATIONS:
Overall Officials: David A Scheiner, MD, Principal Investigator — University Hospital of Zurich, Clinic for Gynaecology
Locations (1):
- University Hospital of Zurich, Clinic for Gynaecology, Zurich, Switzerland